CLINICAL TRIAL: NCT05684900
Title: Research of the Effect of Reservoir Oxygen Mask Application on Respiratory and Hemodynamic Parameters in Sedated Adult Patients for Gastrointestinal System Endoscopy
Brief Title: Research of the Effect of Reservoir Oxygen Mask Application on Respiratory Parameters in Sedated Adult Patients for Gastrointestinal System Endoscopy
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aydoğan Çelik, MD,Anesthesiology and Reanimation, Derince Training and Research Hospital
Other Study IDs: DERINCETRHCELIK001
Record Dates: First submitted 2022-11-29; First posted 2023-01-13 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- reservoir oxygen mask: During the sedation procedure in the endoscopy unit, patients who used a reservoir oxygen mask will be examined. No premedication will be applied to patients admitted to the endoscopy unit. As a standard, intravenous vascular access will be established with a 22 gauge intraket on the back of the left hand in all patients, 6-10 lt/minute oxygen therapy will be started with a reservoir mask, and peripheral oxygen saturation, end-tidal CO2, blood pressure arterial values will be monitored and recorded. These parameters will be monitored and recorded every five minutes during the procedure. In addition, the sedative agents applied to the patients and their doses will be recorded. After the procedure, all patients will be taken to the recovery room, where they will be observed until the modified aldrete score is 9 or higher. The recovery times of the patients, nausea, vomiting and similar symptoms will be followed and recorded.

SUMMARY:
With the oxygen mask with reservoir, oxygen can be given to patients with FiO2 values that can reach 80-100%. Reservoir oxygen mask is superior to other oxygen treatment methods with the high oxygen rate applied.Our hypothesis is that the use of an oxygen mask with a reservoir will reduce the incidence of respiratory complications in adult patients who will undergo sedation in the endoscopy unit.

DETAILED DESCRIPTION:
During the sedation procedure in the endoscopy unit, patients who used a reservoir oxygen mask will be examined. Patients over the age of 18 and under the age of 70, with ASA 1-2 risk score, who are planned to be operated under sedation in the endoscopy unit of our hospital will be included. Patients who do not have verbal and written consent to participate in the study, have an ASA3-4 risk score, and are scheduled for emergency procedures will be excluded from the study. No premedication will be applied to patients admitted to the endoscopy unit. As a standard, intravenous vascular access will be established with a 22 gauge intraket on the back of the left hand in all patients, 6-10 lt/minute oxygen therapy will be started with a reservoir mask, and peripheral oxygen saturation, end-tidal CO2, blood pressure arterial values will be monitored and recorded. These parameters will be monitored and recorded every five minutes during the procedure. In addition, the sedative agents applied to the patients and their doses will be recorded. After the procedure, all patients will be taken to the recovery room, where they will be observed until the modified aldrete score is 9 or higher. The recovery times of the patients, nausea, vomiting and similar symptoms will be followed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and under the age of 70
* Patienst with have an ASA1-2 risk score

Exclusion Criteria:

* Patients who do not have verbal and written consent to participate in the study
* Patienst with have an ASA3-4 risk score,
* Patients scheduled for emergency intervention.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who used an oxygen mask with a reservoir during the sedation procedure in the endoscopy unit will be examined.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Post-anaesthetic discharge scoring criteria | up to 2 HOUR
  In the modified aldrete scoring system, 5 criteria such as activity, respiration, circulation, consciousness and oxygen saturation are evaluated.Patients with a modified Aldrete score of 9 and above can be sent to the service.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydoğan Çelik, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided